CLINICAL TRIAL: NCT01267110
Title: Engaging Diverse Underserved Communities to Bridge the Mammography Divide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Kimberly Engelman, PhD, Associate Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 12371
Record Dates: First submitted 2010-12-21; First posted 2010-12-24 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: MI2 intervention arm
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: MI2 intervention arm — For persons who are randomized to the MI2 intervention arm, the HLK-BH program will guide participants through a series of questions to fully delineate step-by-step breast cancer screening intentions of participants the when, where and how of screening)and encourage follow through on these intentions.
  Arms: Intervention
Other: Control — Each participant in the C intervention arm will receive the same brief one-on-one breast cancer screening education information delivered in person by a CHW as MI2 participants. In additional participants will go through the Healthy Living Kansas-Breast Health computerized screening and intervention program.
  Arms: Control

SUMMARY:
Breast cancer is the second most common cause of cancer death in the U.S.1 in spite of being preventable, easily detectable, and curable.2-11 Breast screening continues to be underutilized by the general population and especially by traditionally underserved minority populations. Two of the least screened minority groups are American Indians/Alaska Natives (AI/AN) and Latinas. American Indian/Alaska Native women have the poorest recorded 5-year cancer survival rates of any ethnic group and the lowest (or near-lowest) screening rates for major cancers.12 Furthermore, breast cancer is the number one cause of cancer mortality among Latina women.13 While breast cancer screening rates have increased nationally, there has been an increase in the gap in breast cancer screening utilization between individuals from minority versus majority racial/ethnic groups.

DETAILED DESCRIPTION:
If you decide to participate in the program, your participation will last 4 months. You will complete the Healthy Living Kansas-Breast Health survey by computer. The survey will take about 20 minutes to complete. You will be randomly assigned (like flipping a coin) to one of two groups. The groups will receive different breast health information. After completing the survey, you agree to be contacted by telephone in 4 months to answer questions. You will be asked for your name, home address, and phone number.

You will be given information about breast cancer and mammography. You may or may not benefit from the information provided. Care will be taken to safeguard the information you provide but under rare circumstances confidentiality breaches may occur.

ELIGIBILITY:
Inclusion Criteria:

* Latina or AI/AN woman residing in one of participating communities
* Aged ≥40 years of age
* Not up to date on mammography screening
* Home address & access to a working telephone
* Responded to 120-day post randomization follow-up call

Exclusion Criteria:

* Receipt of mammogram within past year
* Acute medical illness, history of breast cancer, 1st
* Cognitive impairment or inappropriate affect or behavior
* Another household member enrolled in the study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-09; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
120-day post randomization mammography screening completion | day 120
  To compare the 120-day post randomization mammography screening completion rates of individuals who receive a computerized mammography "implementation intentions" (MI2) intervention, versus a comparison computerized condition of general breast cancer prevention health education (C).

SECONDARY OUTCOMES:
To compare the screening mammography self-reported barriers after 120-days post randomization | day 120
  To compare the screening mammography self-reported barriers after 120-days post randomization between those receiving a mammography "implementation intentions" intervention (MI2) and those receiving only a general breast cancer prevention health education intervention (C).
To compare changes in mammography screening Precaution Adoption Process Model | day 120
  To compare changes in mammography screening Precaution Adoption Process Model decisional stage from baseline to 120 days post randomization between individuals in the MI2 and C study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Engelman, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Engelman KK, Cupertino AP, Daley CM, Long T, Cully A, Mayo MS, Ellerbeck EF, Geana MV, Greiner A. Engaging diverse underserved communities to bridge the mammography divide. BMC Public Health. 2011 Jan 21;11:47. doi: 10.1186/1471-2458-11-47. PMID 21255424